CLINICAL TRIAL: NCT00308048
Title: 14 vs 24 Weeks HCV Treatment to Genotype 2/3 Patients With Rapid Virological Response
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ullevaal University Hospital (Other)
Collaborators: Schering-Plough (Industry)
Organization: Oslo University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P03720
Record Dates: First submitted 2006-03-27; First posted 2006-03-28 (Estimated); Last update posted 2011-07-06 (Estimated); Status verified 2006-03

CONDITIONS: Hepatitis C Virus Infection
Keywords: Interferon; Pegylated interferon; Pegylated interferon alfa 2b; Hepatitis C; Genotype 2; Genotype 3; Rapid virological response; Short treatment; 14 weeks treatment; health related quality of life; sick leave; Injecting drug use
MeSH Terms: conditions — Hepatitis C | interventions — Ribavirin

INTERVENTIONS:
Drug: Pegylated Interferon alfa 2b and ribavirin

SUMMARY:
Patients with HCV genotype 2 or 3 infection who have a rapid virological response to treatment are randomised to either 14 or 24 weeks HCV treatment. Our hypothesis is that there is no important difference in effect between the two treatment effect.

DETAILED DESCRIPTION:
Patients with HCV genotype 2 or 3 infection are currently recommended 6 months treatment with pegylated interferon alfa (2a or 2b) and ribavirin.Approximately 80% obtain sustained virological response (HCV RNA undetectable 6 months after treatment) to this approach. However, the treatment is associated with many and sometimes serious side effects. In addition, the treatment is costly also in econimical terms. Increasing the treatment duration beyond 6 months does not increase the response rate. Shorter treatment has only been assessed in small trials, but the results have been encouraging.

In this randomised, open label,multicenter phase 3 trial with acitive controls patients are treated with pegylated interferon alfa 2a (PegIntron (R), Schering Plough NJ)(1,5 mcg/kg)and ribavirin (Rebetol (R), Schering Plough, NJ) (800-1400mg based on weight)for 4 weeks. Those who are HCV RNA negative at week 4 (<50 IU; Cobas Amplicor Monitor Test, Roche Diagnostic) are defined as rapid virological responders and randomised to either an additional 10 or 20 weeks combination treatment. Patients who are HCV RNA positive are all treated for 20 more weeks. The endpoint is sustained virological response defined as undetectable HCV RNA 24 weeks after end of treatment.

Our hypothesis is that there is no important difference in the effect in the two groups.

This is a non-inferiority trial. The smallest difference considered to be clinically important is 10%. Thus to state "non-inferiority" the 95% confidence interval of the observed difference between the groups shall not overlap 10%. Both intention to treat and and per protocol analyses will be published. Conclusion will be conservative and based on the analysis who detect the biggest difference.

ELIGIBILITY:
Inclusion Criteria:

HCV RNA positive Genotype 2 or 3 Treatment naive Raised ALT

-

Exclusion Criteria:

Active substance abuse Poorly controlled psychiatric disease Decompensated cirrhosis HBsAg positive Anti-HIV positive Suffering from other significant concurrent medical conditions including chronic liver diseases -

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 435
Dates: Start 2004-03; Study Completion 2006-09

PRIMARY OUTCOMES:
Sustained virological response (SVR) =HCV RNA negativity (<20 IU/ml) six months after end of treatment.

SECONDARY OUTCOMES:
Change in health related quality as measured by short from 36 (SF-36) from baseline to 6 months after end of treatment.
Sick leave in patients treated for 14 or 24 weeks treatment

CONTACTS AND LOCATIONS:
Overall Officials: Olav Dalgard, MD PhD, Principal Investigator — Ullevaal University Hospital, Oslo, Norway
Locations (1):
- Ullevaal University Hospital, Oslo, Norway

REFERENCES:
- [Background] Dalgard O, Bjoro K, Hellum KB, Myrvang B, Ritland S, Skaug K, Raknerud N, Bell H. Treatment with pegylated interferon and ribavarin in HCV infection with genotype 2 or 3 for 14 weeks: a pilot study. Hepatology. 2004 Dec;40(6):1260-5. doi: 10.1002/hep.20467. PMID 15558712